CLINICAL TRIAL: NCT06658535
Title: Novel Oxygen Therapeutic NanO2 for Mild Respiratory Distress in Phase 1b
Brief Title: A Dose Escalation Study of NanO2 in Patients With Mild Respiratory Distress
Acronym: EXTEND-1b
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NuvOx LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EXTEND 1b; 75A50123C00034 (Other Grant/Funding Number: ASPR-BARDA)
Record Dates: First submitted 2024-09-26; First posted 2024-10-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Mild Respiratory Distress
Keywords: respiratory distress
MeSH Terms: conditions — Dyspnea | interventions — perfluoropentane

STUDY DESIGN:
Intervention Model Description: Up to six subjects will be enrolled at each dose level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 0.025 (Experimental): Loading dose = 0.025 mL/kg followed sustained IV infusion of 0.375 mL/kg over 21 hours.
  Interventions: Drug: dodecafluoropentane (0.025 mL/kg)
- Cohort 0.032 (Experimental): Loading dose of 0.032 mL/kg followed sustained IV infusion of 0.48 mL/kg over 21 hours.
  Interventions: Drug: dodecafluoropentane (0.032 mL/kg)
- Cohort 0.050 (Experimental): Loading dose of 0.050 mL/kg followed by sustained IV infusion of 0.75 mL/kg over 21 hours.
  Interventions: Drug: dodecafluoropentane (0.050 mL/kg)

INTERVENTIONS:
Drug: dodecafluoropentane (0.025 mL/kg) — dodecafluoropentane (0.025 mL/kg)
  Other Names: NanO2™
  Arms: Cohort 0.025
Drug: dodecafluoropentane (0.032 mL/kg) — dodecafluoropentane (0.032 mL/kg)
  Other Names: NanO2™
  Arms: Cohort 0.032
Drug: dodecafluoropentane (0.050 mL/kg) — dodecafluoropentane (0.050 mL/kg)
  Other Names: NanO2™
  Arms: Cohort 0.050

SUMMARY:
EXTEND is a dose escalation study of NanO2™ in patients with mild respiratory distress who are at risk for mechanical ventilation. The study will establish dosing guidelines for a Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* Requiring supplemental oxygen but ≤ 6L oxygen by nasal cannula to maintain an oxygen saturation >92% or PaO2 >60mmHg
* Admitted to a hospital with symptoms of mild RD
* Signed informed consent obtained from the subject or subject's legally authorized representative
* Agrees to not participate in another clinical trial for the treatment of mild RD through Day 28

Exclusion Criteria:

* Presence of extracorporeal membrane oxygenation
* Unstable hypertension
* History of significantly impaired renal function defined as an eGFR ≤ 30mL/min/1.73m2 (MDRD equation or similar) or impaired hepatic function defined as the presence of decompensated cirrhosis (acute deterioration in liver function characterized by jaundice, ascites, hepatic encephalopathy, hepatorenal syndrome, or variceal hemorrhage)
* Presence of pulmonary embolism at baseline
* Evidence of right ventricular heart failure
* Unstable hemodynamically as defined by receiving 0.5μg/kg/min or greater norepinephrine
* Inability to comply with the study procedures
* Currently pregnant or breastfeeding
* Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 48 hours
* History or evidence of any other clinically significant condition that, in the opinion of the investigator, might pose a safety risk to subjects or interfere with study procedures, evaluation, or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 28 Days
  To determine the Maximum Tolerated Dose of NanO2 in subjects with Mild Respiratory Distress.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 days
  Cumulative incidence of adverse events and serious adverse events

OTHER OUTCOMES:
Change in Respiratory Rate Oxygenation (ROX) Index score | 24 hours
  Change in ROX Index from baseline. ROX Index = 100*(SaO2/FiO2)/respiratory rate
World Health Organization (WHO) 8-point scale for clinical assessments | 28 days
  Evaluate distribution of WHO 8-point ordinal scale at various time points throughout the study. Clinical assessment assigning clinical status of increasing severity from 1 to 8.
NanO2 Oxygenation | 2 days
  Duration of NanO2 oxygenation response as measured by pulse oximetry
Determine the effects of NanO2 on PaO2 measurements | 2 days
  Comparisons of PaO2 measurements before, during and after NanO2 infusions

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Grey Nun Community Hospital, Edmonton, Alberta
  - Hôpital Maisonneuve Rosemont, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided